CLINICAL TRIAL: NCT05923385
Title: Are Static and Dynamic Balance Tests A Criteria Showing Cognitive Impairments In the Elderly?
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, Prof.Dr., Biruni University
Other Study IDs: Biruni Univers
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Geriatric Population; Balance Problems
Keywords: geriatria; cognitive status; balance test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Four Square Step Test — These are standardized test which will be applied to subjects with pencil, paper and time recorder.
  Other Names: Timed Get Up and Go Test; One Leg Standing Test (Eyes Open and Eyes Closed); Standardized Mini Mental Test; Functional Reach Test

SUMMARY:
The aim of our study is to reveal whether static and dynamic balance tests can be an indicator of deterioration in cognitive impairments in geriatric individuals.

DETAILED DESCRIPTION:
the static and dynamic balance test will be used to predict cognitive impairments in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Relative, healthy elderly individuals aged 65-85 years
* Individuals who do not have neurological / orthopedic problems that will prevent them from performing the test
* Independent elderly individuals in activities of daily living
* Men and women living in a nursing home
* No pre-defined vision and hearing problems
* No history of lower extremity or lumbar spinal surgery

Exclusion Criteria:

* Hadkinson's Abbreviated Mental Test less than 7 points
* Presence of defined neurological, orthopedic, systemic (cardiovascular) disease that interferes with walking and mobility
* Presence of defined psychiatric illness
* Having a communication problem
* Presence of using aids for walking
* Use of prostheses or orthoses associated with the lower extremity
* Presence of cognitive, visual or auditory impairment
* Balance-affected individuals with lower extremity disorders

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Relative healthy nursing home residents aged 65-85 living in the nursing home will be included in the study.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | 5 minutes
  The mini mental test is a test that can be administered by a physician, nurse, psychologist or a healthcare professional with a short training. It is a practical mental test in terms of applicability that can show the cognitive level globally. Evaluates cognitive performance quantitatively. It is important in terms of examining the course of dementia cases and their response to treatment in the clinic. There are 11 items in the test gathered around 5 main headings. These items are; Orientation is register memory, attention and calculation, recall and language. The total score is evaluated out of 30. A score of 25 and above is considered normal. Between 10 and 19 is moderate dementia. Between 19-24 refers to early dementia (13,14).
Four Step Square Test | 8 minutes
  The test clinically assesses the ability to change direction while taking a step. At the start of the test, the patient stands in the upper left square (Frame 1) and looks in the direction of Square 2. First, the step sequence is clockwise: Square 1, then Squares 2, 4, and 3. Then the step sequence is counterclockwise: square 3, followed by squares 4, 2, and 1. The physiotherapist demonstrates the test and allows the patient to apply the model to learn the sequence. The test is repeated if the patient fails to complete the sequence successfully or loses balance or touches the cane. Two points are obtained and the better of these two points is recorded. Timed effort begins when the first foot touches the ground at Square 2 and then ends when the patient's second foot touches the ground at Square 1 (15, 16, 17).
Timed Up and Get Test | 5 minutes
  The test assesses functional mobility, balance, and performance in adults 65 years and older. Wearing normal shoes and walking aids, the patient begins the test in a standard seat with his back against the chair, his arms resting on the arms of the chair, and both feet flat on the floor. The patient is instructed to stand up and walk to a line on the ground at a distance of 3 m, turn on the line, walk back to the chair and sit on the chair. The test ends when the patient's hip touches the seat.
  The test is repeated twice; The fastest time is recorded. It is classified as mobile for <10 s, general independent for <20 s, and limited mobility for >30 s (15, 16, 18).

SECONDARY OUTCOMES:
One Leg Standing Test (Eyes Open and Eyes Closed): | 3 minutes
  One leg is lifted without touching the standing leg. Initially, the eyes remain open. The patient is instructed to close their eyes and is asked to maintain their balance for 30 seconds. Balance disorder is suspected if the lifted leg touches the support leg, the lifted leg touches the ground, the patient jumps on the standing leg, or touches something for balance. Inability to balance on one leg for 30 seconds during one-leg stance is an indication of decreased balance function. However, the clinical expectation for the ability to balance on one leg decreases with the age of the patient. Healthy individuals aged 60-69 should be able to stand on one leg with their eyes open for at least 5 seconds (19).
Functional Reach Test: | 4 minutes
  The functional reach test, developed by Duncan et al., is a reliable and validated test used in clinical balance measurement. Have the patient raise the right arm 90° while standing in a comfortable position with bare feet and then step with the right arm without stepping and/his balance. During the functional reach test, the physiotherapist observes whether the patient is on the ground with both feet and does not step forward. If one of these behaviors occurs, the patient repeats the test. The Functional Reach Test is repeated three times and the best measurement is recorded. Decreased ability to lie down indicates an increased risk of the patient falling in the future; Values of 15 cm and below indicate a significantly increased risk of falling, and values between 15 and 25 cm indicate a mild fall risk (20).

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, PT,PhD., Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Thapa PB, Gideon P, Fought RL, Kormicki M, Ray WA. Comparison of clinical and biomechanical measures of balance and mobility in elderly nursing home residents. J Am Geriatr Soc. 1994 May;42(5):493-500. doi: 10.1111/j.1532-5415.1994.tb04970.x. PMID 8176143
- [Background] Leipzig RM, Cumming RG, Tinetti ME. Drugs and falls in older people: a systematic review and meta-analysis: II. Cardiac and analgesic drugs. J Am Geriatr Soc. 1999 Jan;47(1):40-50. doi: 10.1111/j.1532-5415.1999.tb01899.x. PMID 9920228
- [Background] Boyd R, Stevens JA. Falls and fear of falling: burden, beliefs and behaviours. Age Ageing. 2009 Jul;38(4):423-8. doi: 10.1093/ageing/afp053. Epub 2009 May 6. PMID 19420144
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Duncan RP, Earhart GM. Four square step test performance in people with Parkinson disease. J Neurol Phys Ther. 2013 Mar;37(1):2-8. doi: 10.1097/NPT.0b013e31827f0d7a. PMID 23364168
- [Background] Shubert TE, McCulloch K, Hartman M, Giuliani CA. The effect of an exercise-based balance intervention on physical and cognitive performance for older adults: a pilot study. J Geriatr Phys Ther. 2010 Oct-Dec;33(4):157-64. PMID 21717919
- [Background] Gunendi Z, Ozyemisci-Taskiran O, Demirsoy N. The effect of 4-week aerobic exercise program on postural balance in postmenopausal women with osteoporosis. Rheumatol Int. 2008 Oct;28(12):1217-22. doi: 10.1007/s00296-008-0651-3. Epub 2008 Jul 22. PMID 18648815
- [Background] Harrison JK, McArthur KS, Quinn TJ. Assessment scales in stroke: clinimetric and clinical considerations. Clin Interv Aging. 2013;8:201-11. doi: 10.2147/CIA.S32405. Epub 2013 Feb 18. PMID 23440256
- [Background] Stevenson TJ, Garland SJ. Standing balance during internally produced perturbations in subjects with hemiplegia: validation of the balance scale. Arch Phys Med Rehabil. 1996 Jul;77(7):656-62. doi: 10.1016/s0003-9993(96)90004-0. PMID 8669991
- [Background] Schulz BW, Hart-Hughes S, Gordon MT, Bulat T. Training implications of maximal forces on a computer-controlled and motor-driven leg press by age group, sex, footplate direction, and speed. Exp Gerontol. 2012 Apr;47(4):295-303. doi: 10.1016/j.exger.2012.01.003. Epub 2012 Jan 20. PMID 22289381